CLINICAL TRIAL: NCT06565637
Title: Targeting Minority Stressors to Improve Eating Disorder Symptoms in Sexual Minority Individuals With Eating Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Tiffany Brown, Assistant Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R61MH133710-01A; 1R61MH133710-01 (NIH)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Eating Disorders; Sexual Minorities
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psychotherapy (Experimental): Participants in this arm will experience the PRIDE intervention. PRIDE is a 14-session treatment that incorporates aspects of cognitive behavioral therapy for eating disorders (CBT-E) and SM-affirmative therapy. CBT-E aspects of treatment include in-session weighing, self-monitoring (food logs), regular eating, and techniques to address overvaluation of weight and shape. SM-affirmative therapy techniques include discussing the impact of minority stress on health, resilience, and strength within the SM community, specific manifestations of minority stress on eating and body image, current coping strategies, emotion regulation skills, and developing mindful, present-focused reactions to minority stress.
  Interventions: Behavioral: Promoting Resilience to Improve Disordered Eating

INTERVENTIONS:
Behavioral: Promoting Resilience to Improve Disordered Eating — See description under "Arms"
  Other Names: PRIDE

SUMMARY:
The goal of this clinical trial is to learn if a new intervention (Promoting Resilience to Improve Disordered Eating; PRIDE) can decrease internalized stigma and increase the ability to cope effectively with stressors in sexual minority populations diagnosed with eating disorders. The main question it aims to answer is:

Will an eating disorders treatment focused on decreasing internalized stigma and increasing sexual minority stress coping self efficacy in sexual minority populations? Participants Will

* Complete a telephone screen with study staff to determine preliminary eligibility for the study
* Undergo a behavioral eligibility screening that includes structured clinical interviewing in order to determine proper diagnosis of an eating disorder along with ensuring absence of non-eating disorder diagnoses
* Complete self-report measures to determine study eligibility
* Attend up to 14 weekly therapy sessions as part of the PRIDE intervention, where participants will work with qualified clinicians to address eating pathology and disordered body image along with developing effective strategies for coping with sexual minority stressors
* Complete surveys upon completion of the intervention 3 and 6 months post follow-up

DETAILED DESCRIPTION:
Eating disorders are one of the deadliest psychiatric disorders and are associated with high economic burden (over $65 billion annually in the United States), and numerous physical health consequences. One of the most at-risk groups for developing eating disorders are sexual minority (SM; e.g., gay, lesbian, bisexual, pansexual, queer, non-heterosexual) individuals. Indeed, existing research finds that SM individuals have a 2-3 fold risk for developing an eating disorder compared to their non-SM peers and the these disparities have persisted during the past decade, with no signs of attenuating. This increased risk is due, in part, to chronic stressors (e.g., prejudice, victimization, discrimination) and subsequent SM stress reactions (e.g., internalized stigma) due to being part of a marginalized group. SM individuals experiencing perceived discrimination for their SM identity are 5-times more likely to develop an eating disorder. Data, including those from a large sample across the United States support that, in particular, internalized stigma is associated with increased eating disorder symptom severity in SM men and women. Prior research also supports in the face of SM stressors, SM individuals may be more likely to use maladaptive coping strategies, leading to low SM-stress coping self-efficacy, which has subsequently been shown to lead to disordered eating.

Despite this inequity, there are no known eating disorder treatments developed specifically for SM individuals to address the distinct processes that increase and maintain eating disorder risk. Further, existing treatments for eating disorders are only effective for ~50% of patients, calling for more targeted approaches. SM adults have been accessing eating disorder treatment at increasing rates over the last decade. However, pilot data from our group also suggests that SM individuals are also more likely to drop out of eating disorder treatment compared to their non-SM peers, suggesting that culturally sensitive treatments to address the unique needs of SM individuals with eating disorders are needed. To address this gap, and consistent with a mechanism-informed experimental therapeutics approach, the proposed study will test an innovative, virtually-delivered, treatment (Promoting Resilience to Improve Disordered Eating; PRIDE) integrating current evidence-based treatment for eating disorders with techniques and principles of SM-affirmative treatment to address SM stressors that are posited to maintain eating disorder symptoms. If PRIDE exerts a clinically meaningful effect on the posited targets (i.e., internalized stigma, SM-stress coping self-efficacy) during the R61 phase in a sample of n = 30 participants and is feasible/acceptable, the investigators will move to the R33 phase.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* identify as lesbian, gay, bisexual, other non-heterosexual identities
* meet criteria for a Diagnostic and Statistical Manual - 5 (DSM-5) eating disorder (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder, other specified feeding or eating disorder)
* reports current (past 12 months) experience with discrimination due to sexual orientation;
* speaks English
* has internet access and a working webcam
* reside (and plan to continue to reside for the study duration) in California or one of the Psychology Interjurisdictional Compact (PSYPACT) states
* able to provide informed consent

Exclusion Criteria:

* inability to speak/read English
* active suicidal plans or intent
* other major untreated psychiatric diagnoses (e.g., untreated bipolar disorder, untreated psychosis)
* body mass index below 17.0, a standard clinical cutoff used to denote moderate-severe underweight that may be indicated for a higher level of medical care than standard outpatient treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Internalized Homophobia Scale (IHP) | Change from Baseline through 3- and 6-month follow-up
  Assesses internalized stigma (9 items, 5-point scale, higher scores indicate greater internalized stigma).
Sexual Orientation Implicit Association Test | Change from Baseline through 3- and 6-month follow-up
  Assesses internalized stigma via computerized behavioral task involving categorizing positive/negative words with sexual minority and heterosexual people.
Coping Self Efficacy Scale (CSES) | Change from Baseline through 3- and 6-month follow-up
  Assesses sexual minority(SM)-stress coping self efficacy, as adapted for address SM stress in prior research (13 items, 11-point scale, higher scores indicate greater SM-stress coping self-efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Brown, PhD, Principal Investigator — Auburn University; Aaron Blashill, PhD, Principal Investigator — San Diego State University
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - San Diego State University, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
Data will be available via NDA in compliance with the National Institute of Mental Health (NIMH) grant funding. Researchers will be able to use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable. As an alternative, instructions for contacting investigators (MPIs) will be placed on their lab websites so that researchers interested in using the data can contact them directly to obtain the de-identified data. The research team will require that any recipients of the data execute a data sharing agreement with Auburn University that will obligate recipients to 1) use data only for research; 2) not identify an individual participant; 3) commit to securing data using appropriate computer technology; and 4) commit to destroying or returning data after analyses are completed or three years have passed.